CLINICAL TRIAL: NCT02820857
Title: Assessment of the Efficacy of Bevacizumab in Combination With Folfiri as Second-line Treatment After the Failure of the Cisplatin (or Carboplatin)-Etoposide Combination in Patients Suffering From an Advanced Inoperable Poorly Differentiated Neuroendocrine Carcinoma of an Unknown or Gastroentero-pancreatic Primary Cancer. A Phase 2 Non-comparative Randomized Study
Brief Title: Assessment of the Efficacy of Bevacizumab in Combination With Folfiri as Second-line Treatment in Patients Suffering From an Advanced Inoperable Poorly Differentiated Neuroendocrine Carcinoma of an Unknown or Gastroentero-pancreatic Primary Cancer
Acronym: BEVANEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL14_0442; 2016-001305-16 (EudraCT Number)
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Neuroendocrine Carcinomas
Keywords: Gastroentero-pancreatic neuroendocrine carcinomas; Second-line treatment; Bevacizumab; Folfiri
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Folfiri-bevacizumab (Experimental): Patient treated with a combination Folfiri-bevacizumab. Treatment every 2 weeks (D1 = D15)
  Interventions: Drug: Folfiri-bevacizumab
- Folfiri (Active Comparator): Patient treated with Folfiri only. Treatment every 2 weeks (D1 = D15)
  Interventions: Drug: Folfiri

INTERVENTIONS:
Drug: Folfiri-bevacizumab — Patient treated with a combination Folfiri-bevacizumab. Treatment every 2 weeks (D1 = D15)
  Arms: Folfiri-bevacizumab
Drug: Folfiri — Patient treated with Folfiri only. Treatment every 2 weeks (D1 = D15)
  Arms: Folfiri

SUMMARY:
Poorly differentiated neuroendocrine carcinomas (NEC) are a sub-group of aggressive neuroendocrine neoplasms (NEN). The most common primary sites are broncho-pulmonary and digestive. The gastroentero-pancreatic NECs (GEP-NEC) represent 7-21% of all of the NENs.

Recent data on the initial presentation of GEP-NEC have been reported in two retrospective studies and a French cohort study. No standard second-line treatment has been defined for NECs. Despite a very negative prognosis, these NECs have a certain amount of chemosensitivity, close to that of bronchial NECs. Multiple-drug therapies such as Folfiri, or Folfox, or single drug treatments such as temozolomide are the proposed options but with a low level of proof Bevacizumab associated with a cytotoxic chemotherapy has shown promising results in well differentiated neuroendocrine tumors (NET), known for being hypervascular. The efficacy of bevacizumab has also been suggested in patients with NEC, but never in the context of a phase II study. Its combination with Folfiri is efficient and well tolerated in metastatic colorectal cancer. The combination Folfiri-bevacizumab potentially represents an optimized treatment compared to chemotherapy with only Folfiri. No phase II or III studies have reported results for these patients, and no on-going phase II or III trial have been identified to date.

The main objective of this study is to show that, after the failure of a first-line chemotherapy using platinum-etoposide, the combination Folfiri-bevacizumab allows significant prolongation of overall survival in adult patients with GEP-NEC.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged ≥ 18 years old,
* Poorly differentiated neuroendocrine carcinoma (NEC) from a gastrointestinal tract (from esophagus to anal canal) and biliopancreatic primary or an unknown primary cancer, locally advanced and/or metastatic,
* Centralized review of the diagnostic by a consulting pathologist specializing in NET (TENPATH network),
* Recommendation of a second-line chemotherapy after progression, documented using the RECIST criteria v.1.1, and after a first-line chemotherapy treatment by cisplatin (or carboplatin) + etoposide or in the event of progression in the 6 months following the discontinuation of this first-line treatment,
* Recommendation of a second-line chemotherapy for the refractory patient or contraindicated for platinum-etoposide chemotherapy
* Patients presenting at least one measurable target lesion according to the RECIST criteria v.1.1, in an area not previously irradiated,
* General condition ≤ 2 (WHO),
* Patient of child bearing age accepting to use an effective contraception during treatment and until 6 months after the last administration,
* Patient who signed the informed consent form.

Exclusion Criteria:

1. Relating to the tumor, the patient, and previous treatment:

   * Well differentiated neuroendocrine tumor
   * Mixed tumor, except if the NEC component is > 70%, the patient is eligible,
   * First-line chemotherapy other than cisplatin (or carboplatin) and etoposide,
   * All malignant disease in the three years before randomization, with the exception of basal cell carcinoma or in situ cancer treated for curative purposes,
   * A pregnant or breastfeeding woman,
   * Lack of efficient contraception (for men or women of reproductive age),
   * All medical, geographical, social, and psychological conditions or a legal situation that will not allow the patient to finish the study or sign an informed consent form,
2. Relating to the chemotherapy (Folfiri):

   * Any of the following uncontrolled progressive diseases in the 6 months before randomization: liver failure, renal insufficiency, respiratory distress, congestive heart failure (NYHA III-IV), unstable angina, myocardial infarction, significant arrhythmia,
   * Known deficiency in dihydropyrimidine dehydrogenase,
   * Known Gilbert's syndrome,
   * Total bilirubin level >1.5x the upper limit of normal (ULN); AST (Aspartate transaminase) and/or ALT (Alanine transaminase) >5x ULN; TP <50%;
   * Neutrophils <1.5x109/l, platelets <100x109/l, hemoglobin <9 g/dl,
   * Chronic uncontrolled diarrhea, unresolved intestinal occlusion or subocclusion,
   * History of anaphylactic reaction or known intolerance to atropine (sulfate) or to loperamide or to antiemetics administered in association with Folfiri,
   * All treatment with concomitant anticonvulsive agents, CYP3A4 inducers (phenytoin, phenobarbital, carbamazepine), discontinued for at least 7 days,
3. Relating to bevacizumab:

   * Uncontrolled brain metastases (by local treatment),
   * All uncontrolled progressive disease within 1 month prior to randomization: grade 3-4 gastrointestinal bleeding (peptic ulcer, erosive esophagitis or gastritis), infectious disease or intestinal inflammation, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event,
   * Uncontrolled high blood pressure defined as a systolic blood pressure >140 mmHg or diastolic pressure >90 mmHg,
   * Patients receiving anticoagulant treatment with an unstable dose of a vitamin K antagonist treatment, and/or having an abnormal INR (>3) in the four weeks before the randomization,
   * Verified proteinuria above or equal to 1g/24 hours measured from 24 hours of urine if the urinary protein dipstick control is above or equal to 2+,
   * Creatinine clearance (MDRD) <50 ml/min.
   * Hypersensitivity to the active substance or to any of the excipients.
   * Hypersensitivity to Chinese Hamster Ovary (CHO) cell products or other recombinant human or humanised antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
Proportion of patients alive | 6 months after treatment
  The primary endpoint is the proportion of patients alive 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (26):
- France (26):
  - Service d'Hépato-Gastroenterologie et Oncologie Digestive, Hôpital Sud, CHU d'Amiens, Amiens
  - Service d'Hépatogastroentérologie, CHU d'Angers, Angers
  - Service d'Oncologie et Radiothérapie, Institut Sainte Catherine, Avignon
  - Service de Gastroentérologie et Oncologie Digestive, Hôpital Avicenne, Bobigny
  - Service de Gastroentérologie et Pancréatologie, Hôpital Beaujon, APHP, Clichy
  - Service de Gastroentérologie, CHU Henri Mondor, Créteil
  - Service d'Hépato-Gastroentérologie et Oncologie Digestive, CHU de Dijon, Dijon
  - Service d'Hépatogastroentéologie, Hôpital Michallon, CHU de Grenoble, Grenoble
  - Département de Cancérologie Urologique et Digestive, Centre Oscar Lambret, Lille
  - Département de cancérologie médicale - Groupe des tumeurs endocrines, Centre Léon Bérard, Lyon
  - Service d'Oncologie Médicale - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - Département d'Oncologie Médicale, Institut Paoli Calmettes, Marseille
  - Service d'Hépato-Gastroentérologie et d'Oncologie Digestive, Hôpital de la Timone, APHM, Marseille
  - Service d'Oncologie Médicale, Hôpital Saint Eloi, CHU de Montpellier, Montpellier
  - Service d'Hépatogastroentérologie, CHR d'Orléans, Orléans
  - Département d'Oncologie Médicale, Hôpital Saint-Antoine, Paris
  - Service de Gastroentérologie, Hôpital Cochin, APHP, Paris
  - Service d'Hépato-Gastroenterologie et Oncologie Digestive, Hôpital Européen Georges Pompidou, APHP, Paris
  - Service d'Hépato-Gastroentérologie et d'Oncologie Digestive, Hôpital Haut Lévêque, CHU Bordeaux, Pessac
  - Pôle Régional de Cancérologie, CHU de Poitiers, Poitiers
  - Service d'Hépato-Gastroentérologie et Cancérologie, Hôpital Robert Debré, CHU de Reims, Reims
  - Service d'Hépatogastroentérologie, Hôpital Pontchaillou, CHU de Rennes, Rennes
  - Service de Gastroentérologie, CHU de Rouen, Rouen
  - Service de Gastro-Entérologie, Hôpital Nord, CHU de ST-Etienne, Saint-Priest-en-Jarez
  - Service d'Oncologie Médicale, Hôpital Civil, CHU de Strasbourg, Strasbourg
  - Service d'Oncologie Endocrinienne, Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walter T, Lievre A, Coriat R, Malka D, Elhajbi F, Di Fiore F, Hentic O, Smith D, Hautefeuille V, Roquin G, Perrier M, Dahan L, Granger V, Sobhani I, Mineur L, Niccoli P, Assenat E, Scoazec JY, Le Malicot K, Lepage C, Lombard-Bohas C. Bevacizumab plus FOLFIRI after failure of platinum-etoposide first-line chemotherapy in patients with advanced neuroendocrine carcinoma (PRODIGE 41-BEVANEC): a randomised, multicentre, non-comparative, open-label, phase 2 trial. Lancet Oncol. 2023 Mar;24(3):297-306. doi: 10.1016/S1470-2045(23)00001-3. Epub 2023 Feb 2. PMID 36739879